CLINICAL TRIAL: NCT07068373
Title: Development of Evidence Based Therapeutic Guidelines for Early Speech and Language Acquisition in Urdu Speaking Children With Cochlear Implant
Brief Title: Development of Evidence-based Therapeutic Guidelines for Early SLA in Urdu-speaking Children With Cochlear Implants
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: PhDRSW/Batch-Fall23/2225
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mixed method (Exploratory Sequential) — 4-6 Expert SLPs working with Cochlear Implant, A cohort of 100 Urdu speaking children who received cochlear implants

SUMMARY:
Firstly global and regional literature on speech therapy after cochlear implantation focusing on Urdu-speaking populations and culturally relevant factors will be systematically reviewed.

DETAILED DESCRIPTION:
Then needs Assessment will be done to understand the challenges, needs, and gaps in therapeutic practices specific to Urdu-speaking children through focus groups to gather insights into current practices and barriers. After that objective data will be collected to identify trends and outcomes in speech and language development post-implantation, measure baseline skills, and progress over time, and factors influencing outcomes i.e. age of implantation, therapy frequency. In final stage, culturally relevant and evidence-based therapeutic guidelines will be formulated.

ELIGIBILITY:
Inclusion Criteria:

* Speech language Pathologists/ therapist with minimum 5 years of experience working with cochlear implant
* Parents of children with cochlear implant age 2 and above

Exclusion Criteria:

* Parents whose children has just cochlear implant and they have no experience of speech and language development after cochlear implant

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Early Speech and Language acquisition of Urdu speaking children after cochlear implant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Likert scale | 18 Months
  A Likert scale is a psychometric scale commonly used in questionnaires to measure respondents' attitudes and opinions. It typically presents a statement and asks respondents to indicate their level of agreement or disagreement using a range of ordered response options. These options are usually assigned numerical values for scoring purposes. Scoring is designed based on such categories as "Strongly Disagree," "Disagree," "Neither Agree nor Disagree," "Agree," and "Strongly Agree." (0-5) for each question, the higher the score indicates the worse condition

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore City, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No